CLINICAL TRIAL: NCT06679569
Title: Effect of Deep Neuromuscular Blockade on Postoperative Pain in Pediatric Patients Undergoing Laparoscopic Surgery: a Prospective Randomized Controlled Trial
Brief Title: Deep Neuromuscular Blockade on Postoperative Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ji-Hyun Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2410-015-1575
Record Dates: First submitted 2024-11-04; First posted 2024-11-07 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- moderate neuromuscular blockade (Active Comparator)
  Interventions: Drug: rocuronium 0.2 mg/kg/hr continuous infusion
- deep neuromuscular blockade (Experimental)
  Interventions: Drug: rocuronium 0.6 mg/kg/hr continuous infusion

INTERVENTIONS:
Drug: rocuronium 0.2 mg/kg/hr continuous infusion — To maintain Train-of-four count 1 to 3 during surgery: Administration of continuous infusion of rocuronium at a rate of 0.2 mg/kg/hr to achieve and sustain moderate neuromuscular blockade.
  Arms: moderate neuromuscular blockade
Drug: rocuronium 0.6 mg/kg/hr continuous infusion — To maintain Train-of-four count 0 during surgery: Administration of continuous infusion of rocuronium at a rate of 0.6 mg/kg/hr to achieve and sustain deep neuromuscular blockade.
  Arms: deep neuromuscular blockade

SUMMARY:
This study aims to investigate the impact of varying degrees of neuromuscular blockade on postoperative pain in pediatric patients aged over 2 months to under 7 years undergoing laparoscopic surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged over 2 months to under 7 years scheduled for laparoscopic surgery under general anesthesia.
* American Society of Anesthesiologists (ASA) Physical Status Classification I, II, or III.

Exclusion Criteria:

* Patients undergoing emergency surgery.
* Patients with chronic pain or currently taking analgesics for chronic pain.
* Known hypersensitivity to general anesthetic agents or analgesics.
* Patients with underlying cardiovascular disease.
* Patients with neuromuscular disorders.
* Any other condition that, in the investigator's judgment, would make the patient unsuitable for participation in the study.

Ages: 2 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-11-06 (Estimated); Study Completion 2026-11-07 (Estimated)

PRIMARY OUTCOMES:
ANIm (Analgesia Nociception Index) Value | 30 minutes after arrival in the recovery room

SECONDARY OUTCOMES:
FLACC Pain Scale | 30 minutes after arrival in the recovery room
Pediatric Anesthesia Emergence Delirium Scale | 30 minutes after arrival in the recovery room
Time to Extubation | From end of surgery to extubation (in minutes, assessed up to 1 hour)
Recovery Room Length of Stay | Duration of stay in the recovery room (in minutes, assessed up to 2 hours)
Remifentanil Consumption During Anesthesia | During surgery ( assessed up to 5 hours)
  mcg/kg/min
Change in Pain Score (FLACC Pain Scale) | Every 6 hours up to 24 hours post-surgery
Maximum Pain Score (FLACC Pain Scale) within 24 Hours | Within 24 hours post-surgery
Total Narcotic/Non-Narcotic Analgesic Consumption per Body Weight | Within 24 hours post-surgery
Peak Intraabdominal Pressure During Surgery | During surgery (assessed up to 5 hours)
Peak Inspiratory Pressure During Surgery | During surgery (assessed up to 5 hours)
Leiden Surgical Rating Scale | During surgery (assessed up to 5 hours)
Events During Recovery (Agitation, Stridor, Desaturation < 95%, Nausea, Vomiting, Bradycardia, Oxygen Requirement) | During recovery room stay (assessed up to 2 hours)
Any complications Occurring Before Discharge | Up to discharge (assessed up to 1 month)

CONTACTS AND LOCATIONS:
Locations (1):
- SNUCH, Seoul, Seoul, South Korea